CLINICAL TRIAL: NCT02877602
Title: Patient Understanding of LiverMultiScan
Status: Completed | Type: Observational
Sponsor: Perspectum (Industry)
Responsible Party: Sponsor
Other Study IDs: Patient LMS
Record Dates: First submitted 2016-08-17; First posted 2016-08-24 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Experience of liver disease: This is defined as either those who have had direct experience of liver disease as sufferers, or the carers of those who have had liver disease. Each individual receives an MRI (LiverMultiScan), with many also receiving a FibroScan.
  Interventions: Device: MRI; Device: Transient Elastography

INTERVENTIONS:
Device: MRI
  Other Names: LiverMultiScan
Device: Transient Elastography
  Other Names: FibroScan

SUMMARY:
This is a qualitative study to determine which factors affect the patient experience of having a liver MRI, what information patients would like to receive after their MRI, and how patients would like this information communicated to them.

DETAILED DESCRIPTION:
This is a qualitative study to determine which factors affect the patient experience of having a liver MRI, what information patients would like to receive after their MRI, and how patients would like this information communicated to them. Each individual will receive at least an MRI scan (LiverMultiScan), with many also receiving a FibroScan (Transient Elastography). Patients will then undergo a focused qualitative interview, as well as filling out a questionnaire. The interviews will be thematically analysed and trends identified by significance.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with experience of liver disease.
* Individuals over the age of 16.
* Individuals willing to give informed consent for participation in the study.

Exclusion Criteria:

* Individuals with any contraindication to magnetic resonance imaging.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with experience of liver disease, either as a sufferer or carer.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Factors effecting MRI experience and understanding. | Immediately (within 1 hour) after undergoing the MRI scan, and receiving results feedback.
  This will be analysed based on themes and trends emanating from answers within the focused interview and questionnaire following the scan, and results feedback.

SECONDARY OUTCOMES:
Comparison of MRI to ultrasound scan in terms of patient experience. | Immediately (within 1 hour) after undergoing an MRI scan, and ultrasound (FibroScan) scan.
  This will be analysed based on themes and trends emanating from answers within the focused interview and questionnaire following the scan, and results feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Rajarshi Banerjee, BM BCh MRCP MSc DPhil, Principal Investigator — Perspectum Diagnostics
Locations (1):
- University of Oxford Centre for Clinical Magnetic Resonance Research (OCMR), Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McKay A, Pantoja C, Hall R, Matthews S, Spalding P, Banerjee R. Patient understanding and experience of non-invasive imaging diagnostic techniques and the liver patient pathway. J Patient Rep Outcomes. 2021 Sep 10;5(1):89. doi: 10.1186/s41687-021-00363-5. PMID 34508298